CLINICAL TRIAL: NCT01488721
Title: Clinical Evaluation of the xMAP® NeoPlex4™ Assay for Detection of T4, TSH, 17-OHP and IRT Using the NeoPlex System
Brief Title: Clinical Evaluation of NeoPlex4 Assay and NeoPlex System
Status: Completed | Type: Observational
Sponsor: Luminex Corporation (Industry)
Responsible Party: Sponsor
Organization: Luminex Molecular Diagnostics (Industry)
Other Study IDs: CLD-0001
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Adrenal Hyperplasia, Congenital; Congenital Hypothyroidism; Cystic Fibrosis
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Congenital Hypothyroidism; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- General Newborn Population-Prospective: Specimens prospectively collected in the course of routine newborn screening originating from hospitals, birthing centers, and/or clinics.
- Newborn Specimens-Confirmed Positive: Banked confirmed positive specimens that were originally collected as part of the newborn screening program, but when found to screen positive for a disease, were followed up clinically to definitively diagnose the subject with the disease (CF, CAH or CH). Follow up results were reported to the sites by the treating clinicians.

SUMMARY:
The purpose of this study is to assess the agreement of clinical performance between the proposed NeoPlex 4 assay and NeoPlex System and the comparator devices in clinical use in newborn screening programs for detection of T4, TSH, 17-OHP and IRT.

DETAILED DESCRIPTION:
The proposed (investigational) NeoPlex4 assay measures levels of thyroxine (T4), thyrotropin (hTSH), 17-alpha-OH-progesterone (17-OHP) and immunoreactive trypsinogen (IRT) from dried blood specimens (DBS) collected from neonates to screen for congenital hypothyroidism (CH), congenital adrenal hyperplasia (CAH) and cystic fibrosis (CF). The Clinical Evaluation of the xMAP® NeoPlex4™ Assay (NeoPlex4) for Detection of T4, TSH, 17-OHP and IRT using the NeoPlex System is a multi-center method concordance study on a combination of prospectively collected neonatal dried blood spots and pre-selected archived frozen dried blood spots that have been demonstrated to be positive for 17-OHP (CAH), IRT (CF), and T4 or TSH (CH). The study will be conducted at selected sites that routinely perform newborn screening testing in the United States.

ELIGIBILITY:
Inclusion Criteria:

* The dried blood spot specimen was collected on an FDA-cleared collection paper that has not yet passed its expiration dating.
* Prospective specimens used in this study should only be those collected for the first time from a subject, or initial collection specimens.

Exclusion Criteria:

* Collected within 24 hours of birth.
* Specimens stored at ambient temperature for greater than 14 days prior to testing.
* The specimen DBS appears diluted.
* The specimen DBS shows evidence of clotting, caking, layering or serum rings.
* The DBS punched disks were punched too close to the edge of the blood spot or show printed markings.
* The specimen or collection card was contaminated with fecal material.
* Non-eluting blood spot due to deterioration of sample caused by exposure to heat and humidity.

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Specimens will be derived from prospectively collected neonatal specimens and banked neonatal specimens originating from hospitals, birthing centers, and/or clinics. Newborn screening is currently performed on all neonates; there is no selection criterion for subjects.
Sampling Method: Probability Sample
Enrollment: 7462 (Actual)
Dates: Start 2011-12; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Smith, PhD, Study Director — Luminex Corporation
Locations (3):
- United States (3):
  - New York State Department of Health, Albany, New York
  - Tennessee Department of Health, Nashville, Tennessee
  - Unified State Laboratories: Public Health, Taylorsville, Utah